CLINICAL TRIAL: NCT06837415
Title: Association Between Preoperative Anxiety and Blood Eosinophil Levels; a Prospective Study.
Brief Title: Association Between Preoperative Anxiety and Blood Eosinophil Levels
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2019.04.98
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Anxiety; Preoperative Evaluation; STAI; Eosinophil Blood Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — complete blood count, blood eosinophil count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm control
- Arm eosinophilia

SUMMARY:
In the studies, the presence of preoperative anxiety has been evaluated and reported with anxiety scales. The presence of anxiety and allergic diseases has also been examined in a limited study with the analysis of neuroendocrine cells. In this study, it was planned to support the eosinophilia response in peripheral blood accelerated by stress-related anxiety with anxiety scales. In patients who apply to the anesthesia clinic before surgery, the preoperative anxiety level will be measured with the STAIT(The State-Trait Anxiety Inventory Test) and APAIS (The Amsterdam Preoperative Anxiety and Information Scale) scales performed before the anesthesia evaluation and the relationship with the eosinophil count in the patient's complete blood count analysis will be evaluated.

DETAILED DESCRIPTION:
Anxiety is an unpleasant emotion that affects patient comfort. Surgery is a significant trauma and is significantly associated with patient anxiety. Postoperative pain expectations, separation from family, inadequacy, loss of independence, and fear of surgery and death increase perioperative anxiety symptoms. Therefore, preoperative anxiety has the potential to change the dynamics of an elective surgical procedure. If mismanaged, it can lead to postponement or cancellation of surgical procedures. Both outcomes have clinical and economic detrimental effects. Studies on patients undergoing elective surgery have shown that anxiety, depression, somatoform disorder, and fear of pain are frequently encountered, while the prevalence of preoperative anxiety varies between 11% and 80%, and is an important factor that increases perioperative morbidity in adults. Several factors have been associated with preoperative anxiety. These factors include low education level, female gender, age, type of surgery, marital status, social status, ASA grade, psychiatric illness, previous poor clinical experiences, specific types of surgery, smoking, and BMI. In practice, many documents have been reported in the evaluation of preoperative anxiety, and the most commonly used test is the STAI scale. In addition, the APAIS, which is simpler and less time-consuming to administer, was developed to measure anxiety and desire for information related to anesthesia and surgery, and its usability and correlation with the STAI were investigated.

Recently, a few studies have shown a relationship between anxiety and allergic diseases. The relationship between allergic symptoms and psychological disorders is complex. Chronic allergy, especially asthma, is a source of psychological distress in itself. On the other hand, dysfunctional psychological reactions have a negative effect on the perception and management of allergy symptoms. Side effects such as fatigue, weakness, joint pain, swelling, headache and psychological disorders usually accompany allergies and greatly impair the quality of life of patients. It has been reported that there is a relationship between allergy and psychological dysfunction, namely anxiety, depression and decreased ability to cope with stress, and that the frequency of anxiety in allergic patients is as high as 19%. Atopic predisposition is defined as a personal or family history of type 1 allergy, bronchial asthma, allergic rhinitis and conjunctivitis and/or atopic dermatitis and/or a tendency to overproduction of IgE (immunoglobulin E) antibodies. Some anxiety disorders have been detected in 35% of 100 cases of type I atopy. It has been shown that atopic patients have high anxiety levels, both in children and adults, and that psychotherapy improves not only the psychological but also the dermatological condition. Different studies have focused on the importance of mental stress as a cause of atopic dermatitis or asthma exacerbations in children and adults. Although the effect of stress on skin lesions is not fully understood, recent studies have shown that it both mediates anxiety and affects immune function. Acute psychological stress leads to an increase in the number of eosinophils in the peripheral blood of patients with atopic dermatitis. Eosinophilia is characterized by an increase in the number of complete peripheral eosinophils. It has three categories: mild (500-1500 /mm3), moderate (1500-5000/mm3) and severe (>5000/mm3). The clinical effect of eosinophilia is variable. Based on studies, the limit blood eosinophil value defining patients with eosinophilic asthma has been shown as 0.3 x 109 L -1. While a significant advantage in preventing exacerbations has been reported in patients with eosinophil count <150, this advantage has not been identified in cases where the whole blood eosinophil count is >150.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery
* Have sufficient language skills for the interview
* Ages 16-85
* ASA I - III
* Patients who apply to the anesthesia clinic for anesthesia evaluation

Exclusion Criteria:

* under the age of 16
* Patients who do not consent
* Patients with insufficient language skills
* Patients with mental and/or psychiatric disorders
* Patients with a history of emergency and/or ASA-IV
* sedative drug use

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on patients aged 16-85 years who apply for preoperative anesthesia evaluation for an elective surgical procedure by an anesthesiologist at the Health Sciences University Kanuni Sultan Süleyman E.A.H. Anesthesia Polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood eosinophil count and preoperative anxiety | 1 day (From enrollment to the end of completion of the survey forms)

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)